CLINICAL TRIAL: NCT03992274
Title: Yunnan-ADARC HIV Prevention Program: Developing and Testing a Model to Implement and Sustain PrEP Delivery in China
Brief Title: Biomedical HIV/AIDS Prevention Program Yunnan
Acronym: B-HAPPY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of support and approval by the Yunnan Provincial Health Authority
Sponsor: Columbia University (Other)
Collaborators: Yunnan Center for Disease Control and Prevention (Other); Oregon Social Learning Center (Other); Hunter College of The City University of New York (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kathrine Meyers, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAS8800; 1R01MH119884-01A1 (NIH)
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: HIV/AIDS
Keywords: HIV prevention; Implementation science; Pre-Exposure Prophylaxis; Men who have sex with men; China
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard implementation (No Intervention): During Standard Implementation, sites will use standard Yunnan Center for Disease Control and Prevention strategies to introduce HIV prevention innovations.
- Enhanced implementation (Experimental): During Enhanced Implementation, sites will transition to receive enhanced Implementation Support to plan and implement PrEP.
  Interventions: Other: Enhanced implementation of PrEP

INTERVENTIONS:
Other: Enhanced implementation of PrEP — During Enhanced Implementation study sites will receive Implementation Support to plan and introduce PrEP by following the eight stages of the PrEP-adapted SIC. Implementation Support specifically will involve a centralized technical assistance system developed using US-based PrEP experience focused on addressing implementation issues identified through real-time analysis of client, clinic, and implementation data.
  Arms: Enhanced implementation

SUMMARY:
B-HAPPY is an implementation project to study the process by which pre-exposure prophylaxis (PrEP) is introduced and integrated into a specific international health system facing high rates of HIV incidence among men who have sex with men. The study will use a stepped wedge design to compare implementation outcomes across eight municipalities in Yunnan, China.

DETAILED DESCRIPTION:
B-HAPPY is an implementation science project that will introduce and evaluate the implementation of PrEP among over 1000 men who have sex with men (MSM), in eight municipalities in Yunnan, China. The project aims to compare the effectiveness of two implementation strategy bundles: 1) Standard Implementation: comprising the strategies that the Yunnan Center for Disease Control and Prevention would usually use to introduce HIV prevention innovations in the absence of the proposed study; and 2) Enhanced Implementation: standard implementation enhanced by a SIC-guided approach to plan and implement PrEP.

This study will use a stepped-wedge design, where sites will go through four study periods: a Pre-Baseline Period (Routine Service with no PrEP Implementation), a Baseline Period (Standard Implementation of PrEP), an Experiment Period (Enhanced Implementation of PrEP), and a Post-Experiment-Observation Period. Sites are randomized to the timing of the intervention initiation, with 2 sites moving from Standard Implementation to Enhanced Implementation every 6 months. The intervention condition changes over time and the intervention effect is the difference in outcomes between the Baseline and Experiment Periods, and the Post-Experiment and Baseline Periods.

The specific aims of the proposed study are:

1. To evaluate whether the addition of SIC-guided PrEP delivery (Enhanced Implementation) to standard health system PrEP delivery improves services outcomes. Through a stepped-wedge randomized trial across eight Yunnan municipalities, within site change over time will be examined; timing of introduction of Enhanced Implementation will be randomized across four cohorts of two sites each. Client-services outcomes include progress to achieving the "Five-80s" (patient PrEP awareness, screening, offering, initiation, continuation).
2. To examine the implementation process and efficiency of the Enhanced versus Standard implementation approaches. Using the Stages of Implementation Completion (SIC) and Cost of Implementing New Strategies (COINS) tools, sites will be monitored for implementation process and resource use. Outcomes will include proportion of implementation activities completed; duration of each implementation phase; and cost and resource allocation for completion of each implementation phase.

ELIGIBILITY:
This study will recruit two types of study participants: A. MSM clients at study sites; B. study staff who will be involved in the implementation of this project.

A. MSM clients:

Inclusion criteria:

Clients at study sites (VCT or STI [sexually transmitted infections] clinics) are eligible for inclusion in the study if they meet all of the following criteria:

* Aged 18 years or older
* Male sex at birth
* Willing and able to provide written consent form
* Able and willing to provide finger-scan and contact information
* Not infected with HIV-1
* Any male sex partner in past 12 months

Exclusion Criteria:

Clients at study sites (VCT or STI clinics) will be excluded from the study if they meet any of the following criteria:

* Diagnosed with HIV or AIDS
* Signs or symptoms of acute HIV infection
* Unable to provide inform consent
* At enrollment, has any medical, psychological, or social condition that, in the opinion of the investigator, would jeopardize the health or wellbeing of the participant during the study or the integrity of the data

B. Study staff:

Inclusion criteria:

Staff at study sites (VCT or STI clinics) are eligible for inclusion in the study if they meet all of the following criteria:

* Aged 18 years or older
* Employed at site for at least 3 months
* Willing and able to provide consent

Exclusion criteria:

Staff at study sites (VCT or STI clinics) will be excluded from the study if they meet any of the following criteria:

* Unable to provide consent
* At enrollment, has any medical, psychological, or social condition that, in the opinion of the investigator, would jeopardize the health or wellbeing of the participant during the study or the integrity of the data

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathrine Meyers, DrPH,MPP,MSc, Principal Investigator — Aaron Diamond AIDS Research Center, Columbia University
Locations (1):
- Yunnan Center for Disease Prevention and Control, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
Data from the B-HAPPY project will be available at end of the project by contacting the study PI.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants include clients and staff. The study was conducted at 8 study sites Yunnan, China.
Pre-assignment Details: No participants or sites progressed beyond the Pre-Baseline.
Units Other Than Participants: sites
Groups:
- Sequence 1: 6 Months Pre-Baseline, Then 6 Months Baseline: Sequence 1: 6 months Pre-Baseline, 6 months Standard Implementation, 12 months Enhanced Implementation, and 6 months Post-Experiment Observation.
  Pre-Baseline: Routine Service with no PrEP Implementation.
  Baseline Period: Standard Implementation of PrEP.
  Experiment Period: Enhanced Implementation of PrEP.
- Sequence 2: 6 Months Pre-Baseline, Then 12 Months Baseline: Sequence 2: 6 months Pre-Baseline, 6 months Standard Implementation, 12 months Enhanced Implementation, and 6 months Post-Experiment Observation
  Pre-Baseline: Routine Service with no PrEP Implementation.
  Baseline Period: Standard Implementation of PrEP.
  Experiment Period: Enhanced Implementation of PrEP.
- Sequence 3: 6 Months Pre-Baseline, Then 18 Months Baseline: Sequence 3: 6 months Pre-Baseline, 18 months Standard Implementation, 12 months Enhanced Implementation, and 6 months Post-Experiment Observation
  Pre-Baseline: Routine Service with no PrEP Implementation.
  Baseline Period: Standard Implementation of PrEP.
  Experiment Period: Enhanced Implementation of PrEP.
- Sequence 4: 6 Months Pre-Baseline, Then 24 Months Baseline: Sequence 4: 6 months Pre-Baseline, 24 months Standard Implementation, 12 months Enhanced Implementation, and 6 months Post-Experiment Observation
  Pre-Baseline: Routine Service with no PrEP Implementation.
  Baseline Period: Standard Implementation of PrEP.
  Experiment Period: Enhanced Implementation of PrEP.
Period: Overall Study
Arm/Group | Sequence 1: 6 Months Pre-Baseline, Then 6 Months Baseline | Sequence 2: 6 Months Pre-Baseline, Then 12 Months Baseline | Sequence 3: 6 Months Pre-Baseline, Then 18 Months Baseline | Sequence 4: 6 Months Pre-Baseline, Then 24 Months Baseline
Started | 114; 8 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites
Clients | 58; 8 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites
Staff | 56; 8 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites
Completed | 114; 8 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites
Not Completed | 0; 0 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites

BASELINE CHARACTERISTICS:
Groups:
- Clients: MSM clients (men who have sex with men) who are involved in PrEP implementation
- Staff: Program staff who are involved in PrEP implementation
- Total: Total of all reporting groups
Arm/Group | Clients | Staff | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Customized [Count of Participants; unit: Participants]
  >=18 years old | 58 | 56 | 114
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/Gender data were not collected from staff.
  Participants
    number analyzed (Participants) | 58 | 0 | 58
    Female | 0 |  | 0
    Male | 58 |  | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 58 | 56 | 114
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 58 | 56 | 114
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 58 | 56 | 114

OUTCOME MEASURES:

1. Primary Outcome: PrEP Awareness
Description: Number of clients who are aware of PrEP
Time Frame: Up to 48 months
Population: Due to the closure of the study and loss of funding, intervention was not implemented, and data was not collected or analyzed.
Groups:
- Standard and Enhanced Implementation: The participants would be randomized into Standard OR Enhanced Implementation groupings. However, because the study was stopped early, the participants had not yet been randomized.
  During Standard Implementation, sites will use standard Yunnan Center for Disease Control and Prevention strategies to introduce HIV prevention innovations.
  During Enhanced Implementation, sites will transition to receive enhanced Implementation Support to plan and implement PrEP.
Arm/Group | Standard and Enhanced Implementation
Number analyzed (Participants) | 0

2. Primary Outcome: PrEP Eligible
Description: Number of clients who are eligible for PrEP
Time Frame: Up to 48 months
Population: as for outcome 1
Arm/Group | Standard and Enhanced Implementation
Number analyzed (Participants) | 0

3. Primary Outcome: PrEP Offer
Description: Number of clients who are offered PrEP
Time Frame: Up to 48 months
Population: as for outcome 1
Arm/Group | Standard and Enhanced Implementation
Number analyzed (Participants) | 0

4. Primary Outcome: PrEP Initiation
Description: Number of clients initiating PrEP
Time Frame: Up to 48 months
Population: as for outcome 1
Arm/Group | Standard and Enhanced Implementation
Number analyzed (Participants) | 0

5. Primary Outcome: PrEP Continuation
Description: Number of PrEP initiators who remain PrEP-eligible and sustain use at six months
Time Frame: Up to 48 months
Population: as for outcome 1
Arm/Group | Standard and Enhanced Implementation
Number analyzed (Participants) | 0

6. Primary Outcome: Proportion of PrEP Implementation Activities Completed
Description: The SIC is an 8-stage observational assessment tool recording organizational site completion of implementation activities that map onto the three phases of implementation (Pre-Implementation, Implementation, Sustainability). Proportion of PrEP implementation activities completed will be measured.
Time Frame: Up to 48 months
Population: as for outcome 1
Arm/Group | Standard and Enhanced Implementation
Number analyzed (Participants) | 0

7. Primary Outcome: Time to Completion for Each Implementation Phase
Description: The SIC is an 8-stage observational assessment tool recording organizational site completion of implementation activities that map onto the three phases of implementation (Pre-Implementation, Implementation, Sustainability). Time to completion of each implementation phase will be measured.
Time Frame: Up to 48 months
Population: as for outcome 1
Arm/Group | Standard and Enhanced Implementation
Number analyzed (Participants) | 0

8. Primary Outcome: Cost and Resource Allocation for Completion of Each Implementation Phase
Description: Costs and resource allocation for completion of each implementation phase will be measured with the Cost of Implementing New Strategies (COINS) tool.
Time Frame: Up to 48 months
Population: as for outcome 1
Arm/Group | Standard and Enhanced Implementation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected
Description: Adverse event collection was not done due to study stopping early.
Groups:
- Standard and Enhanced Implementation: During Standard Implementation, sites will use standard Yunnan Center for Disease Control and Prevention strategies to introduce HIV prevention innovations. During Enhanced Implementation, sites will transition to receive enhanced Implementation Support to plan and implement PrEP.
Arm/Group | Standard and Enhanced Implementation
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Due to the lack of support and approval by the Yunnan Provincial Health Authority, the planned study was not able to proceed into the PrEP implementation phase but is considered as completed at the preparatory (pre-baseline) phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT03992274/Prot_SAP_000.pdf